CLINICAL TRIAL: NCT05235438
Title: A Phase 1 Study to Evaluate IMM27M Safety, Tolerability, Pharmacokinetics and Anti-tumor Activity in Patients With Advanced, Metastatic Solid Tumor
Brief Title: Safety and Toxicity Study of IMM27M in Patients With Advanced Solid Tumor
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: ImmuneOnco Biopharmaceuticals (Shanghai) Inc. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IMM27M-001
Record Dates: First submitted 2021-12-22; First posted 2022-02-11 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Oncology; CTLA4 Haploinsufficiency
MeSH Terms: conditions — Neoplasms; Diabetes Mellitus, Insulin-Dependent, 12

STUDY DESIGN:
Intervention Model Description: This study is to observe the dose-limiting toxicity (DLT) of the patients and to determine the maximal tolerance dose(MTD) and recommended dose for expansion (RDE) to observe the AE including relationship and severity of IMM27M based on CTCAE 5.0
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IMM27M (Experimental): IMM27M 0.1, 0.3, 1.0, 2.0, 3.0 mg/kg
  Interventions: Drug: IMM27M

INTERVENTIONS:
Drug: IMM27M — IMM27M injection

SUMMARY:
This is a single arm, open label, multi-center and fist in human dose escalation study, to evaluate the safety, tolerability, pharmacokinetics and anti-tumor activity in patients with advanced and metastatic solid tumor.

DETAILED DESCRIPTION:
Dose escalation (Ia) will recruit 16 disease progress after stand of care(SOC) , no tolerance of SOC solid tumor patients, including malignant melanoma, hepatocellular carcinoma, non-small cell lung cancer, colorectal cancer, ovarian cancer, endometrial cancer, triple negative breast cancer, small cell lung cancer, renal cell carcinoma, squamous cell cancer of head and neck, pancreatic cancer, etc.

IMM27M will be dosed every three weeks (Q3W), the study will be conducted by adjusted 3+3 dose escalation study design, the fist dose is 0.1mg/kg based on the non-clinical study data and NOVEL assessment, the dose level will be 0.1, 0.3, 1.0, 2.0, 3.0 mg/kg, the first dose will recruit 1 patient to avoid patients under no efficacy dose, then the conventional 3+3 study design will start since second dose.

Patients will be observed 3 weeks after the dose, this is also the DLT observation period, patients will be dosed until intolerability, progressed, death or informed consent withdraw, the total duration of treatment will be 48 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Sign an Informed Consent Form voluntarily and comply with the protocol requirements;
2. Age ≥18 years old, and ≤75 years old, regardless of gender;
3. Expected survival ≥12 weeks;
4. Clinical diagnosis:

   Phase Ia: Patients with advanced or recurrent solid tumors diagnosed by histology or cytology, who have previously received standard treatment progress or treatment failure (including progress or relapse after PD-1/PD-L1 inhibitor treatment). Or there is no standard treatment regimen at this stage, including but not limited to malignant melanoma, hepatocellular carcinoma, non-small cell lung cancer, colorectal cancer, ovarian cancer, endometrial cancer, triple negative breast cancer, small cell lung cancer, renal cell carcinoma, squamous cell cancer of head and neck, pancreatic cancer, etc.;
5. Archived tumor histology and pathology reports from fresh or recent treatment can be provided. If tissue specimens are not available, re-biopsy of the tumor is recommended for patients.
6. Lesions can be measured according to the evaluation criteria for solid tumors (RECIST v1.1) (the longest diameter of the spiral CT scan ≥ 10 mm, if the lesion is a lymph node, the short diameter ≥ 15 mm; and radiotherapy has not be performed on the lesion);
7. The performance status ECOG is 0 or 1;
8. For hepatocellular carcinoma (HCC) patients, a Child-Pugh score of A is required, without ascites or hepatic encephalopathy;
9. The organ function level should meet the following requirements:

   Bone marrow: absolute neutrophil count (ANC) ≥1.5×109/L, platelet count ≥85×109/L, hemoglobin ≥90 g/L, and have not received blood transfusion or biological response modifiers (such as granulocyte growth promoting factor, red blood cell growth factor, etc.) ; Note: HCC patients with liver cirrhosis with ANC ≥1.0×109/L and platelet count ≥70×109/L are eligible for enrollment.
   * Liver: total bilirubin (TBIL)≤1.5×ULN, alkaline phosphatase (ALP)≤1.5×ULN, aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5×ULN; if there is liver metastasis, then TBIL≤3.0×ULN, AST and ALT are ≤5.0×ULN; Note: HCC patients with liver cirrhosis with AST and ALT≤5×ULN, TBIL≤3.0×ULN, and albumin ≥2.8g/L are eligible for enrollment.
   * Heart: Left ventricular ejection fraction (LVEF) ≥50% (ECHO confirmed);
   * Kidney: Creatinine (Cr)≤1.5×ULN, or creatinine clearance (Ccr)≥50 mL/min (according to Cockcroft-Gault formula).
   * Thyroid: Thyroid-stimulating hormone (TSH) ≤1×ULN (if abnormal, the levels of FT3 and FT4 should be observed at the same time, if the levels of FT3 and FT4 are normal, they can enroll);
10. Coagulation function: International normalized ratio (INR) ≤ 1.5 × ULN, and activated partial thromboplastin time (APTT) ≤ 1.5 × ULN (except for those who are receiving therapeutic anticoagulant); Note: HCC patients with INR≤2.3×ULN are eligible for enrollment.
11. Adverse events associated with previous systemic chemotherapy, radical/extensive radiotherapy, or other antineoplastic therapy returned to (NCI CTCAE V5.0) ≤ grade 1 (alopecia and peripheral neuropathy < grade 2; except for non-clinical significant or asymptomatic laboratory abnormalities);
12. Patients of childbearing potential should take effective contraceptive during the study to 6 months after the last dose.

Exclusion Criteria:

1. Treatment with the last systemic anti-tumor therapy within 4 weeks prior to the first administration, including chemotherapy, immunotherapy, biotherapy and so on; treatment with hormone anti-tumor therapy and small-molecule targeted therapy within 2 weeks prior to the first administration; palliative local treatment for non-target lesions within 2 weeks prior to the first administration; treatment with non-specific immunomodulatory therapy (such as interleukin, interferon, thymosin, tumor necrosis factor, etc., excluding IL-11 for the treatment of thrombocytopenia) within 2 weeks prior to the first administration; treatment with Chinese herbal medicine or Chinese patent medicine with anti-tumor indications within 1 week prior to the first administration.
2. Treatment with anti-CTLA-4 inhibitors and anti-PD-1/L1 inhibitors 4 weeks before the first administration;
3. Patients with primary central nervous system (CNS) malignant tumors or patients with active metastasis of CNS after local treatment failure (radiotherapy or surgery), but the following patients are allowed to be enrolled: a. Asymptomatic brain metastases; b. Clinical symptoms are stable (i.e., no radiographic progression and all neurological symptoms have returned to baseline 4 weeks before the first administration), and no corticosteroid treatment and other treatments for brain metastasis are required ≥ 4 weeks;
4. Hypertension (systolic blood pressure ≥140mmHg and/or diastolic blood pressure ≥90mmHg), pulmonary hypertension or unstable angina, which cannot be controlled by medication; treatment with myocardial infarction, bypass or stent surgery within 6 months prior to administration; a history of chronic heart failure rated by the New York Heart Association (NYHA) as grade 3-4; valvular disease with clinical significance; severe arrhythmia requiring treatment (excluding atrial fibrillation and paroxysmal supraventricular tachycardia), including QTcF≥450ms for male and ≥470ms for female (calculated by Fridericia formula); cerebrovascular accident (CVA) or transient ischemic attack (TIA) within 12 months prior to enrollment;
5. A history of arterial thrombosis, deep venous thrombosis and pulmonary embolism within 3 months prior to administration;
6. A history of moderate or severe dyspnea at rest due to an advanced malignant tumor or its complications or severe primary pulmonary disease, or a current need for continuous oxygen therapy, or a current history of interstitial lung disease (ILD) or pneumonia, severe chronic obstructive pulmonary disease, severe pulmonary insufficiency, symptomatic bronchospasm, etc.;
7. Development of other malignant tumors within 5 years prior to the first administration. Exceptions: a. Radically cured cervical carcinoma in situ or non-melanoma skin cancer; b. A second primary carcinoma that has been radically cured and has not recurred within 5 years; c. All double primary carcinoma patients can benefit from this study in the opinion of investigators; d. Investigators have definitively excluded what kind of primary tumor the metastasis belongs to;
8. Diseases that may cause gastrointestinal bleeding or perforation (such as duodenal ulcer, intestinal obstruction, acute Crohn's disease, ulcerative colitis, large area gastric and small bowel resection, etc.); patients with chronic Crohn's disease and ulcerative colitis (except for total colon and rectal resection) should be excluded even in inactive phase; patients with hereditary non-polyposis colorectal cancer or familial adenomatous polyposis syndrome; patients with a history of intestinal perforation and intestinal fistula who have not been recovered after surgical treatment; patients with esophageal and gastric varices;
9. Puncture and drainage is needed to treat uncontrollable pleural-peritoneal and pericardial effusions that need repeated drainage or with obvious symptoms;
10. Those with active hepatitis B (HBsAg positive, HBV DNA ≥2000 IU/ml, and excluding hepatitis caused by drugs or other reasons), or active hepatitis C (anti-HCV antibody positive, and HCV RNA higher than lower detection limit);
11. Patients with a history of immunodeficiency, including human immunodeficiency virus (HIV) infection, or other immunodeficiency diseases, or a history of organ transplants;
12. Patients with a history of autoimmune diseases, including but not limited to systemic lupus erythematosus, psoriasis, rheumatoid arthritis, inflammatory bowel disease, Hashimoto's thyroiditis, autoimmune thyroid disease, multiple sclerosis, etc. patient. A history of auto-immune diseases, including but not limited to systemic lupus erythematosus, psoriasis, rheumatoid arthritis, inflammatory bowel disease, Hashimoto's thyroiditis, autoimmune thyroid disorder, multiple sclerosis, etc. Exceptions:

    1. Hypothyroidism that can be controlled by hormone replacement therapy alone;
    2. Dermatosis that does not require systemic therapies (such as vitiligo, psoriasis);
    3. Controlled coeliac disease. Currently under treatment with immunosuppressive agents or systemic hormone therapy (≥10mg/day of prednisone or other hormone equivalents), and still under continued use within 2 weeks prior to enrollment;
13. Evidence of uncontrolled severe active infections (e.g. septicaemia, bacteremia, viremia, etc.);
14. A history of grade 3 or higher allergy (CTCAE v5.0) to any component or excipient of the study drug;
15. Treatment with anti-tumor vaccine therapy or planning to participate in anti-tumor vaccine trials 4 weeks before the first administration;
16. Patients who had major surgery within 4 weeks prior to the first administration and did not recover completely, or who plan to have major surgery in the first 12 weeks after receiving the study drug; patients who had minor surgical procedures (including catheterization, excluding peripherally inserted central catheterization) 2 days before enrollment.
17. Those with a clear history of neurological or mental disorders, such as epilepsy, dementia, and poor compliance;
18. A history of alcohol or drug abuse in the past 1 year;
19. Females who have a positive serum pregnancy test or are breastfeeding; disagree to take adequate contraceptive measures during the study period and 6 months after completion of the study drug;
20. Patients who have participated in other clinical studies in the past shall be out of group in accordance with original clinical studies and more than 4 weeks prior to the first administration of this study;
21. Other situations where investigators believe they are inappropriate for participation in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2022-06-15 (Actual); Primary Completion 2023-08-30 (Estimated); Study Completion 2024-08-30 (Estimated)

PRIMARY OUTCOMES:
a dose-limiting toxicity (DLT) | 3 weeks
  the DLT of IMM27M
The maximum tolerated dose (MTD) and/or recommended dose for expansion (RDE) | 3 weeks
the rate of adverse events | 48 weeks
  the rate of adverse event (AE), severity and relationship of IMM27M based on CTCAE 5.0

SECONDARY OUTCOMES:
Maximum Plasma Concentration (Cmax) | 48 weeks
  the Maximum Plasma Concentration (Cmax) in advanced and relapse patients with IMM27M dosed
Dose escalation: Overall Response Rate (ORR) | 48 weeks
  ORR is defined as the proportion of participants who have a partial response (PR) or better
Dose escalation : Clinical Benefit Rate (CBR) | 48 weeks
  CBR is defined as the proportion of participants who have a critical response (CR), partial response (PR) or disease stable (SD) with at least 12 weeks
Dose escalation : Duration of Response (DOR) | 48 weeks
  DOR is defined as time from date of initial documentation of a response (PR or better) to date of first documented evidence of PD
Dose escalation: Progression-Free Survival (PFS) | 48 weeks
  PFS is defined as time from date of first dose of study drug to date of first documented PD, or death due to any cause, whichever occurs first.
Dose escalation: Disease Control Rate (DCR) | 48 weeks
  DCR is defined as the proportion of participants who have a critical response (CR), partial response (PR) or disease stable (SD)
Incidence of anti-IMM27M | 48 weeks
  To evaluate the immunogenicity of IMM27M in patients with malignancies;
Peak Time (Tmax) | 48 weeks
  the Peak Time (Tmax) in advanced and relapse patients with IMM27M dosed
Area Under the Curve (AUC) | 48 weeks
  the Area Under the Curve (AUC) in advanced and relapse patients with IMM27M dosed
t1/2 | 48 weeks
  the t1/2 in advanced and relapse patients with IMM27M dosed
Plasma clearance (CL) | 48 weeks
  to observe the Plasma clearance (CL) in advanced and relapse patients with IMM27M dosed
Minimum Plasma Concentration (Cmin) | 48 weeks
  the Minimum Plasma Concentration (Cmin) in advanced and relapse patients with IMM27M dosed
Average Plasma Concentration (Cav) | 48 weeks
  the Average Plasma Concentration (Cav) in advanced and relapse patients with IMM27M dosed

CONTACTS AND LOCATIONS:
Locations (6):
- China (6):
  - Peking University First Hospital, Beijing
  - Sun Yai-Sen Memorial Hospital,Sun Yai-Sen University, Guangzhou
  - Sun Yat-sen University Cancer Center, Guangzhou
  - Harbin Medical University Cancer Hospital, Harbin
  - Henan Cancer Hospital, Henan
  - The First Affiliated Hospital of Xi'An Jiaotong University, Xi'an

IPD SHARING:
Plan to Share IPD: No